CLINICAL TRIAL: NCT05675995
Title: Qigong for Post Acute Sequelae of COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Michelle Dossett, Assistant Professor in Residence, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1846783
Record Dates: First submitted 2023-01-04; First posted 2023-01-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Long COVID
Keywords: Qigong
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: Randomized, waitlist controlled design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Receives 6 sessions of qigong first.
  Interventions: Behavioral: Qigong
- Waitlist Control (Other): Receives 6 sessions of qigong after the immediate group
  Interventions: Behavioral: Qigong

INTERVENTIONS:
Behavioral: Qigong — 6 sessions of combined external and internal qigong delivered in a group-based format once a week.

SUMMARY:
The purpose of this study is to conduct a pilot feasibility study of a combination of external and internal qigong on health-related quality of life in individuals with prolonged symptoms following COVID-19 infection.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a combination of external and internal qigong, a traditional Chinese medicine healing practice, improves quality of life and symptoms for individuals with prolonged symptoms following a COVID-19 infection (sometimes called "long COVID"). The study involves completing questionnaires and participating in 6 weekly in person small group qigong sessions with an experienced qigong practitioner.

Participants will be randomized to participate in either an immediate or waitlist control group that will receive the qigong sessions starting 8 weeks later. Participants will complete 3 sets of questionnaires, each about 8 weeks apart and an interview about their experiences with qigong after completing the 6 sessions.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking adults age 18 or greater
2. History of a COVID-19 infection with lingering symptoms lasting longer than 12 weeks
3. Willing and able to access the internet to complete questionnaires
4. Willing and able to travel to the qigong sessions to participate in person in Sacramento, CA.

Exclusion Criteria:

1. Lung scarring secondary to COVID-19 infection as evidenced by signs of parenchymal lung damage on imaging or FVC < 80% (any patient with post COVID-related shortness of breath must have PFTs to be considered for enrollment).
2. Dementia
3. Any other condition that makes it difficult for the individual to complete questionnaires or attend the qigong sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in physical and mental health | 8 weeks
  Changes in PROMIS-29 summary scores from before to after intervention in all participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Must submit written request and complete data sharing agreement.

REFERENCES:
- [Derived] Joy M, Adams N, Yanuck M, Dossett ML. Experiences with Qi and changes in post-acute sequelae of COVID-19 (PASC) symptoms with qigong: a qualitative analysis of participants' experiences in a pilot clinical trial. BMC Complement Med Ther. 2025 Nov 28;25(1):434. doi: 10.1186/s12906-025-05161-w. PMID 41316170